CLINICAL TRIAL: NCT00718718
Title: A Phase 2, 2-Part, Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled, Proof-of-concept, Dose-finding Study Evaluating the Efficacy and Safety of CNTO 136 Administered Subcutaneously in Subjects With Active Rheumatoid Arthritis Despite Methotrexate Therapy
Brief Title: A Study of Effectiveness and Safety of CNTO 136 in Patients With Active Rheumatoid Arthritis Despite Methotrexate Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CR015214; C1377T04 (Other: Centocor); 2007-006603-20 (EudraCT Number)
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Results first posted 2017-12-04 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis, Rheumatoid; Rheumatoid Arthritis; Active Rheumatoid Arthritis; CNTO 136; Interleukin-6; Anti-interleukin-6 monoclonal antibody; Methotrexate; Placebo
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sirukumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (7):
- Part A, Group 1 (Experimental): Participants will receive placebo (Week 0 to Week 10) and later CNTO 136 100 mg (Week 12 to Week 22) every 2 weeks. Stable dose of methotrexate will be maintained through Week 24.
  Interventions: Drug: CNTO 136 100 mg; Drug: Placebo; Drug: Methotrexate
- Part A, Group 2 (Experimental): Participants will receive CNTO 136 100 mg (Week 0 to Week 10) and later placebo (Week 12 to Week 22) every 2 weeks. Stable dose of methotrexate will be maintained through Week 24.
  Interventions: Drug: CNTO 136 100 mg; Drug: Placebo; Drug: Methotrexate
- Part B, Group 1 (Experimental): Participants will receive placebo (Week 0 to Week 10) and later CNTO 136 100 mg (Week 12 to Week 24) every 2 weeks. Stable dose of methotrexate will be maintained through Week 24.
  Interventions: Drug: CNTO 136 100 mg; Drug: Placebo; Drug: Methotrexate
- Part B, Group 2 (Experimental): Participants will receive CNTO 136 100 mg (Week 0 to Week 24) every 2 weeks. Stable dose of methotrexate will be maintained through Week 24.
  Interventions: Drug: CNTO 136 100 mg; Drug: Methotrexate
- Part B, Group 3 (Experimental): Participants will receive CNTO 136 100 mg (Week 0 to Week 24) every 4 weeks and placebo at interim visits (Weeks 2, 6, 10, 14, 18, and 22). Stable dose of methotrexate will be maintained through Week 24.
  Interventions: Drug: CNTO 136 100 mg; Drug: Placebo; Drug: Methotrexate
- Part B, Group 4 (Experimental): Participants will receive CNTO 136 50 mg (Week 0 to Week 24) every 4 weeks and placebo at interim visits (Weeks 2, 6,10, 14, 18, and 22). Stable dose of methotrexate will be maintained through Week 24.
  Interventions: Drug: CNTO 136 50 mg; Drug: Placebo; Drug: Methotrexate
- Part B, Group 5 (Experimental): Participants will receive CNTO 136 25 mg (Week 0 to Week 24) every 4 weeks and placebo at interim visits (Weeks 2, 6,10, 14, 18, and 22). Stable dose of methotrexate will be maintained through Week 24.
  Interventions: Drug: CNTO 136 25 mg; Drug: Placebo; Drug: Methotrexate

INTERVENTIONS:
Drug: CNTO 136 100 mg — CNTO 136 100 mg will be administered subcutaneously (under the skin) every 2 or 4 weeks as per the appropriate randomized arm.
  Other Names: Sirukumab
  Arms: Part A, Group 1; Part A, Group 2; Part B, Group 1; Part B, Group 2; Part B, Group 3
Drug: CNTO 136 50 mg — CNTO 136 50 mg will be administered subcutaneously every 4 weeks from Week 0 to Week 24.
  Other Names: Sirukumab
  Arms: Part B, Group 4
Drug: CNTO 136 25 mg — CNTO 136 25 mg will be administered subcutaneously every 4 weeks from Week 0 to Week 24.
  Other Names: Sirukumab
  Arms: Part B, Group 5
Drug: Placebo — Placebo will be adminstered subcutaneously as per the appropriate randomized arm.
  Arms: Part A, Group 1; Part A, Group 2; Part B, Group 1; Part B, Group 3; Part B, Group 4; Part B, Group 5
Drug: Methotrexate — Stable dose of methotrexate will be maintained through Week 24.

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of subcutaneous (under the skin) administration of anti-interleukin-6 monoclonal antibody (CNTO 136) in reducing signs and symptoms of participants with active rheumatoid arthritis (RA) with methotrexate (MTX) therapy.

DETAILED DESCRIPTION:
This is a multicenter, double-blind (neither physician nor participants knows the treatment that the participant receives), randomized (study medication is assigned by chance), placebo-controlled (an inactive substance is compared with a medication to test whether the medication has a real effect in a clinical study) study. This study will be conducted in 2 parts (Part A and Part B). Each part consists of 3 phases: screening (approximately 1 month prior to the start of study medication), treatment phase (Part A: 22 weeks and Part B: 24 weeks), and follow-up phase (approximately 4 months after the last administration of study medication). In Part A, participants will be randomly assigned to 2 groups to receive CNTO 136 100 mg and placebo for 22 weeks. All participants in Part A, will be crossed over at Week 12 from placebo to CNTO 136 (for Group 1) and from CNTO 136 to placebo (for Group 2). In Part B, participants will be randomly assigned to 5 groups to receive placebo and/or 1 of 3 doses of CNTO 136 (100mg, 50mg or 25mg) for 24 weeks. Participants in Part B, Group 1 will be crossed over at Week 12 from placebo to CNTO 136. All participants should be maintained on a stable dose of MTX for at least 6 weeks prior to the start of study medication through Week 24. Safety will be evaluated by the assessment of adverse events, vital signs, clinical findings, 12-lead electrocardiogram, and clinical laboratory tests which will be monitored throughout the study. The total duration of study participation for a participant will be approximately 42 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with rheumatoid arthritis (RA) for at least 4 months prior to screening
* Have been treated and having an inadequate response with the tolerated dose of methotrexate (MTX) (at least 15mg/week) for at least 4 months prior to screening. MTX doses of 10 or 12.5 mg/week are allowed if participant had intolerance of 15 mg/week
* MTX route of administration and dose (not to exceed 25 mg/week) should be stable for at least 6 weeks prior to the start of the study medication
* Have active RA as defined by persistent disease activity with at least 6 swollen and 6 tender joints, at the time of screening and baseline, and either anti-cyclic citrullinated peptide antibody-positive or rheumatoid factor positive at screening
* C-reactive protein greater than or equal to 1.0 mg/dL (10 mg/L)
* Agree to use one of the contraception methods defined in the protocol

Exclusion Criteria:

* Have inflammatory diseases other than RA that might confound the evaluation of the benefit of CNTO 136 therapy in arthritis
* Family history of/ have long QT syndrome; or a history of second or third-degree heart block
* Received systemic immunosuppressives or disease modifying antirheumatic drug other than MTX, sulfasalazine, hydroxychloroquine or chloroquine within 4 weeks prior to the start of study medication
* Received intra articular (into joints), intramuscular, or intravenous corticosteroids within 4 weeks prior to the start of study medication
* Positive human immunodeficiency virus test, hepatitis B or hepatitis C
* History of / have chronic or recurrent infectious disease, history of / active tuberculosis
* Have serious infection within 2 months prior to start of study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2008-08-11 (Actual); Primary Completion 2011-03-03 (Actual); Study Completion 2011-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor Clinical Trial, Study Director — Centocor, Inc.
Locations (38):
- United States (8):
  - Aventura, Florida
  - Lexington, Kentucky
  - Frederick, Maryland
  - Kalamazoo, Michigan
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Duncansville, Pennsylvania
  - Anderson, South Carolina
- Hungary (3):
  - Budapest
  - Győr
  - Kecskemét
- Japan (8):
  - Goshogawara
  - Hitachi
  - Kawagoe
  - Kitakyushu
  - Miyazaki
  - Sasebo
  - Shinjuku-Ku
  - Tomigusuku
- Mexico (3):
  - Guadalajara
  - Mexico City
  - México
- Poland (8):
  - Bialystok
  - Bydgoszcz
  - Elblag
  - Gdynia
  - Krakow
  - Lublin
  - Poznan
  - Warsaw
- Russia (4):
  - Kemerovo
  - Moscow
  - Novosibirsk
  - Saint Petersburg
- South Korea (4):
  - Busan
  - Daegu
  - Daejeon
  - Seoul

REFERENCES:
- [Derived] Smolen JS, Weinblatt ME, Sheng S, Zhuang Y, Hsu B. Sirukumab, a human anti-interleukin-6 monoclonal antibody: a randomised, 2-part (proof-of-concept and dose-finding), phase II study in patients with active rheumatoid arthritis despite methotrexate therapy. Ann Rheum Dis. 2014 Sep;73(9):1616-25. doi: 10.1136/annrheumdis-2013-205137. Epub 2014 Apr 3. PMID 24699939

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A - Placebo (Wk 0-Wk 12): Participants received placebo subcutaneously (SC) at Week 0 and every 2 weeks (q2w) for 10 weeks.
- Part A - Placebo Then Sirukumab (Wk 12 to End of Study): Participants received 100 mg of sirukumab subcutaneously at Weeks 0, 2 and every 2 weeks (q2w) for Week 10. Thereafter participants received placebo beginning at Weeks 12 and q2w through week 22.
- Part A - Sirukumab (Wk 0-Wk 12): Participants received 100 mg of sirukumab subcutaneously at Weeks 0, 2 and every 2 weeks (q2w) for Week 10.
- Part A - Sirukumab Then Placebo (Wk 12 to End of Study): Participants received placebo at Weeks 12 and q2w through Week 22.
- Part B - Placebo (Wk 0-Wk 12): Participants received placebo subcutaneously (SC) at Week 0 and q2w for 10 weeks.
- Part B - Placebo Then Sirukumab 100 mg q2 Weeks: Participants received placebo subcutaneously (SC) at Week 0 and every 2 weeks (q2w) for 10 weeks. Thereafter participants received sirukumab 100 mg beginning at Weeks 12 and q2w through week 24.
- Part B - Sirukumab 100mg q2w: Participants received 100 mg of sirukumab subcutaneously at Weeks 0, 2 and every 2 weeks (q2w) through Week 24.
- Part B - Sirukumab 100mg q4w: Participants received 100 mg of sirukumab subcutaneously every 4 weeks (q4w) for 24 weeks and in between placebo SC injections was received at Weeks 2, 6, and q4w through week 22.
- Part B - Sirukumab 50mg q4w: Participants received 50 mg of sirukumab subcutaneously every 4 weeks (q4w) for 24 weeks and in between placebo SC injections was received at Weeks 2, 6, and q4w through week 22.
- Part B: Sirukumab 25 mg q4 Weeks: Participants received 25 mg of sirukumabat subcutaneously at Week 0 and every 4 weeks (q4w) for 24 weeks and placebo SC injections at Weeks 2, 6, and q4w through week 22.
Period: Prior to Week 12
Arm/Group | Part A - Placebo (Wk 0-Wk 12) | Part A - Placebo Then Sirukumab (Wk 12 to End of Study) | Part A - Sirukumab (Wk 0-Wk 12) | Part A - Sirukumab Then Placebo (Wk 12 to End of Study) | Part B - Placebo (Wk 0-Wk 12) | Part B - Placebo Then Sirukumab 100 mg q2 Weeks | Part B - Sirukumab 100mg q2w | Part B - Sirukumab 100mg q4w | Part B - Sirukumab 50mg q4w | Part B: Sirukumab 25 mg q4 Weeks
Started | 19 | 0 | 17 | 0 | 30 | 0 | 30 | 30 | 30 | 31
Completed | 18 | 0 | 16 | 0 | 27 | 0 | 29 | 28 | 28 | 31
Not Completed | 1 | 0 | 1 | 0 | 3 | 0 | 1 | 2 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 1 | 0
Not completed — Other | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Week 12 to End of Study
Arm/Group | Part A - Placebo (Wk 0-Wk 12) | Part A - Placebo Then Sirukumab (Wk 12 to End of Study) | Part A - Sirukumab (Wk 0-Wk 12) | Part A - Sirukumab Then Placebo (Wk 12 to End of Study) | Part B - Placebo (Wk 0-Wk 12) | Part B - Placebo Then Sirukumab 100 mg q2 Weeks | Part B - Sirukumab 100mg q2w | Part B - Sirukumab 100mg q4w | Part B - Sirukumab 50mg q4w | Part B: Sirukumab 25 mg q4 Weeks
Started | 0 | 18 | 0 | 16 | 0 | 27 | 29 | 28 | 28 | 31
Treated | 0 | 18 | 0 | 16 | 0 | 26 | 29 | 28 | 28 | 31
Completed | 0 | 17 | 0 | 15 | 0 | 24 | 27 | 27 | 27 | 31
Not Completed | 0 | 1 | 0 | 1 | 0 | 3 | 2 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A: Placebo: Participants received placebo subcutaneously (SC) at Week 0 and every 2 weeks (q2w) for 10 weeks. Thereafter participants received sirukumab 100 mg beginning at Weeks 12 and q2w through week 22.
- Part A: Sirukumab 100 mg q2 Weeks: Participants received 100 mg of sirukumab subcutaneously at Weeks 0, 2 and every 2 weeks (q2w) for Week 10. Thereafter participants received placebo beginning at Week 12 and q2w through week 22.
- Part B: Placebo: Participants received placebo subcutaneously (SC) at Week 0 and every 2 weeks (q2w) for 10 weeks. Thereafter participants received sirukumab 100 milligram (mg) beginning at Week 12 and q2w through week 24.
- Part B: Sirukumab 100 mg q2 Weeks: Participants received 100 mg of sirukumab subcutaneously at Weeks 0, 2 and every 2 weeks (q2w) through Week 24.
- Part B: Sirukumab 100 mg q4 Weeks: Participants received 100 mg of sirukumab subcutaneously at Week 0 and every 4 weeks (q4w) for 24 weeks and placebo SC injections at Weeks 2, 6, and q4w through week 22.
- Part B: Sirukumab 50 mg q4 Weeks: Participants received 50 mg of sirukumab subcutaneously at Week 0 and every 4 weeks (q4w) for 24 weeks and placebo SC injections at Weeks 2, 6, and q4w through week 22.
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A: Sirukumab 100 mg q2 Weeks | Part B: Placebo | Part B: Sirukumab 100 mg q2 Weeks | Part B: Sirukumab 100 mg q4 Weeks | Part B: Sirukumab 50 mg q4 Weeks | Part B: Sirukumab 25 mg q4 Weeks | Total
Number analyzed (Participants) | 19 | 17 | 30 | 30 | 30 | 30 | 31 | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (10.24) | 50.1 (10.72) | 54.1 (12.72) | 53.8 (13.02) | 52 (11) | 50.9 (10.29) | 52.8 (9.41) | 51.8 (11.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25 | 27 | 27 | 26 | 23 | 153
  Male | 8 | 3 | 5 | 3 | 3 | 4 | 8 | 34
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 0 | 0 | 2 | 5 | 3 | 3 | 4 | 17
  Japan | 0 | 0 | 5 | 5 | 5 | 6 | 6 | 27
  Mexico | 0 | 0 | 5 | 3 | 4 | 5 | 6 | 23
  Poland | 13 | 12 | 9 | 10 | 6 | 5 | 7 | 62
  Republic of Korea | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 5
  Russian Federation | 0 | 0 | 9 | 6 | 10 | 9 | 7 | 41
  United States | 6 | 5 | 0 | 0 | 1 | 0 | 0 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 50 Response at Week 12 (Part B)
Description: An American College of Rheumatology (ACR) 50 response is defined as greater than or equal to (>=) 50 percent (%) improvement in both tender joint count (68 joints) and swollen joint count (66 joints) and >= 50% improvement in 3 of the following 5 assessments: participant's assessment of pain using Visual Analogue Scale (Score) VAS (0-10 scale, 0=no pain and 10=worst possible pain), participant's global assessment of disease activity by using VAS (the scale ranges from 0 to 10, [0 = very well to 10 = very poor]), physician's global assessment of disease activity using VAS (the scale ranges from 0 to 10, [0=no arthritis activity to 10=extremely active arthritis]), participant's assessment of physical function as measured by Health Assessment Questionnaire-Disability Index (HAQ-DI, the scale ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area), and serum C-reactive protein (CRP).
Time Frame: Week 12
Population: Population analyzed included all randomized participants in Part B.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part B: Placebo | Part B: Sirukumab 100 mg q2 Weeks | Part B: Sirukumab 100 mg q4 Weeks | Part B: Sirukumab 50 mg q4 Weeks | Part B: Sirukumab 25 mg q4 Weeks
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 31
Percentage of Participants | 3.3 | 26.7 | 23.3 | 26.7 | 19.4
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: Sirukumab 100 mg q2 Weeks; Test type: Superiority or Other; p = 0.026, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: Sirukumab 100 mg q4 Weeks; Test type: Superiority or Other; p = 0.052, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: Sirukumab 50 mg q4 Weeks; Test type: Superiority or Other; p = 0.026, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B: Sirukumab 25 mg q4 Weeks; Test type: Superiority or Other; p = 0.104, Cochran-Mantel-Haenszel

2. Secondary Outcome: Change From Baseline in Disease Activity Index Score 28 (DAS28) Based on C-reactive Protein (CRP) at Week 12 (Part A and Part B)
Description: The DAS28 based on C-Reactive Protein (CRP) is a statistically derived index combining tender joints (28 joints), swollen joints (28 joints), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. The values are 0=best to 10=worst. A negative change from baseline in DAS28 (CRP) (that is, a decrease from baseline) indicates improvement from baseline.
Time Frame: Baseline, Week 12
Population: Population analyzed included randomized subjects in Part A (excluding a site based on sponsor audit for data integrity) and Part B. Here 'n' signifies participants who were evaluable at specific time points, for each arm, respectively.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Part A: Sirukumab 100 mg q2 Weeks: Participants received 100 mg of sirukumab subcutaneously at Weeks 0, 2 and every 2 weeks (q2w) for Week 10. Thereafter participants received placebo beginning at Weeks 12 and q2w through week 22.
Arm/Group | Part A: Placebo | Part A: Sirukumab 100 mg q2 Weeks | Part B: Placebo | Part B: Sirukumab 100 mg q2 Weeks | Part B: Sirukumab 100 mg q4 Weeks | Part B: Sirukumab 50 mg q4 Weeks | Part B: Sirukumab 25 mg q4 Weeks
Number analyzed (Participants) | 19 | 17 | 30 | 30 | 30 | 30 | 31
Units on a Scale
  Baseline: number analyzed (Participants) | 19 | 17 | 29 | 30 | 30 | 29 | 31
  Baseline | 6.341 (0.9034) | 5.919 (0.9676) | 5.908 (0.7332) | 5.755 (0.9706) | 6.190 (0.6829) | 6.051 (0.8791) | 5.688 (0.9529)
  Change at Week 12: number analyzed (Participants) | 17 | 14 | 29 | 30 | 30 | 29 | 31
  Change at Week 12 | -0.619 (0.8541) | -2.075 (0.7979) | -1.073 (0.9766) | -2.248 (1.2050) | -2.011 (0.8843) | -2.198 (0.8550) | -1.964 (0.9532)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Sirukumab 100 mg q2 Weeks; Test type: Superiority or Other; p < 0.001, Van Der Waerden ANOVA
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: Sirukumab 100 mg q2 Weeks; Test type: Superiority or Other; p < 0.001, Van Der Waerden ANOVA
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: Sirukumab 100 mg q4 Weeks; Test type: Superiority or Other; p < 0.001, Van Der Waerden ANOVA
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B: Sirukumab 50 mg q4 Weeks; Test type: Superiority or Other; p < 0.001, Van Der Waerden ANOVA
Statistical Analysis 5: Comparison: Part B: Placebo vs Part B: Sirukumab 25 mg q4 Weeks; Test type: Superiority or Other; p < 0.001, Van Der Waerden ANOVA

3. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 50 Response at Week 12 (Part A)
Description: An ACR 50 response is defined as >= 50% improvement in both tender joint count (68 joints) and swollen joint count (66 joints) and >= 50% improvement in 3 of the following 5 assessments: Participant's assessment of pain using VAS (0-10 scale, 0=no pain and 10=worst possible pain), Participant's global assessment of disease activity by using VAS (the scale ranges from 0 to 10, [0 = very well to 10 = very poor]), Physician's global assessment of disease activity using VAS (the scale ranges from 0 to 10, [0=no arthritis activity to 10=extremely active arthritis]), Participant's assessment of physical function as measured by HAQ-DI (the scale ranges from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area), and Serum CRP.
Time Frame: Week 12
Population: Population analyzed included all randomized participants in Part A (excluding a site based on sponsor audit for data integrity). Here 'N'(number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part A: Placebo | Part A: Sirukumab 100 mg q2 Weeks
Number analyzed (Participants) | 17 | 14
Percentage of Participants | 5.9 | 28.6
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Sirukumab 100 mg q2 Weeks; Test type: Superiority or Other; p = 0.148, Cochran-Mantel-Haenszel

4. Secondary Outcome: Serum Sirukumab Concentrations Through Week 38 (Part A)
Description: Sirukumab Concentrations in serum were measured.
Time Frame: Week 0, Day 2, Day 5, Day 8, Day 11, Week 2, Week 4, Week 8, Week 10, Week 10 Day 4, Week 10 Day 7, Week 12, Week 14, Week 18, Week 22, Week 24, and Week 38
Population: Population analyzed included participants treated with CNTO 136 (Sirukumab) in Part A (excluding a site based on sponsor audit for data integrity). Here 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure whereas 'n' signifies participants evaluable at specific time points, for each arm, respectively.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Part A: Placebo | Part A: Sirukumab 100 mg q2 Weeks
Number analyzed (Participants) | 17 | 14
Microgram per milliliter
  Week 0 | NA (NA) — Data could not be analyzed as the values were below lower limit of quantification (LLOQ) (0.0977 microgram per milliliter). | 0.01 (0.030)
  Day 2: number analyzed (Participants) | 16 | 12
  Day 2 | NA (NA) — Data could not be analyzed as the values were below LLOQ (0.0977 microgram per milliliter). | 3.73 (2.581)
  Day 5: number analyzed (Participants) | 14 | 10
  Day 5 | NA (NA) — Data could not be analyzed as the values were below LLOQ (0.0977 microgram per milliliter). | 7.40 (3.402)
  Day 8: number analyzed (Participants) | 17 | 12
  Day 8 | NA (NA) — Data could not be analyzed as the values were below LLOQ (0.0977 microgram per milliliter). | 6.01 (2.861)
  Day 11: number analyzed (Participants) | 16 | 14
  Day 11 | NA (NA) — Data could not be analyzed as the values were below LLOQ (0.0977 microgram per milliliter). | 5.42 (1.866)
  Week 2: number analyzed (Participants) | 14 | 13
  Week 2 | NA (NA) — Data could not be analyzed as the values were below LLOQ (0.0977 microgram per milliliter). | 4.78 (1.549)
  Week 4: number analyzed (Participants) | 17 | 13
  Week 4 | NA (NA) — Data could not be analyzed as the values were below LLOQ (0.0977 microgram per milliliter). | 8.83 (3.251)
  Week 6: number analyzed (Participants) | 15 | 12
  Week 6 | NA (NA) — Data could not be analyzed as the values were below LLOQ (0.0977 microgram per milliliter). | 10.49 (3.327)
  Week 8: number analyzed (Participants) | 16 | 11
  Week 8 | NA (NA) — Data could not be analyzed as the values were below LLOQ (0.0977 microgram per milliliter). | 12.36 (3.133)
  Week 10: number analyzed (Participants) | 16 | 11
  Week 10 | NA (NA) — Data could not be analyzed as the values were below LLOQ (0.0977 microgram per milliliter). | 13.49 (3.670)
  Week 10 Day 4: number analyzed (Participants) | 12 | 8
  Week 10 Day 4 | NA (NA) — Data could not be analyzed as the values were below LLOQ (0.0977 microgram per milliliter). | 19.07 (4.630)
  Week 10 Day 7: number analyzed (Participants) | 13 | 10
  Week 10 Day 7 | NA (NA) — Data could not be analyzed as the values were below LLOQ (0.0977 microgram per milliliter). | 18.71 (4.111)
  Week 12: number analyzed (Participants) | 12 | 8
  Week 12 | NA (NA) — Data could not be analyzed as the values were below LLOQ (0.0977 microgram per milliliter). | 14.31 (3.438)
  Week 14: number analyzed (Participants) | 16 | 10
  Week 14 | 4.78 (1.779) | 7.07 (2.544)
  Week 18: number analyzed (Participants) | 14 | 9
  Week 18 | 8.52 (4.338) | 2.74 (1.737)
  Week 22: number analyzed (Participants) | 14 | 8
  Week 22 | 10.79 (5.830) | 1.18 (0.816)
  Week 24: number analyzed (Participants) | 13 | 7
  Week 24 | 11.37 (6.177) | 0.88 (0.599)
  Week 38: number analyzed (Participants) | 9 | 6
  Week 38 | 0.41 (0.525) | 0.02 (0.051)

5. Secondary Outcome: Serum Sirukumab Concentrations Through Week 38 (Part B)
Description: Sirukumab Concentrations in serum were measured.
Time Frame: Week 0, Day 5, Day 8, Day 11, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 24 Day4, Week 24 Day7, Week 26, Week 28, Week 30, Week 34 and Week 38
Population: Population analyzed included participants treated with CNTO 136 (Sirukumab) in Part B. Here 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure whereas 'n' signifies participants who were evaluable at specific time points, for each arm, respectively.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Part B: Placebo | Part B: Sirukumab 100 mg q2 Weeks | Part B: Sirukumab 100 mg q4 Weeks | Part B: Sirukumab 50 mg q4 Weeks | Part B: Sirukumab 25 mg q4 Weeks
Number analyzed (Participants) | 26 | 30 | 30 | 30 | 31
Microgram per milliliter
  Week 0: number analyzed (Participants) | 25 | 29 | 30 | 30 | 31
  Week 0 | NA (NA) — Data could not be analyzed as the values were below LLOQ (0.0977 microgram per milliliter). | 0.03 (0.087) | 0.00 (0.000) | 0.02 (0.076) | 0.01 (0.048)
  Day 5: number analyzed (Participants) | 15 | 22 | 22 | 15 | 22
  Day 5 | NA (NA) — Data could not be analyzed as the values were below LLOQ (0.0977 microgram per milliliter). | 6.75 (3.212) | 6.21 (2.933) | 2.66 (1.447) | 1.59 (0.808)
  Day 8: number analyzed (Participants) | 22 | 26 | 28 | 26 | 31
  Day 8 | NA (NA) — Data could not be analyzed as the values were below LLOQ (0.0977 microgram per milliliter). | 5.67 (2.398) | 5.85 (2.774) | 2.61 (1.339) | 1.49 (0.556)
  Day 11: number analyzed (Participants) | 14 | 20 | 18 | 13 | 18
  Day 11 | 0.02 (0.063) | 4.50 (2.307) | 4.68 (2.539) | 2.54 (1.233) | 1.26 (0.516)
  Week 2: number analyzed (Participants) | 20 | 24 | 25 | 25 | 28
  Week 2 | NA (NA) — Data could not be analyzed as the values were below LLOQ (0.0977 microgram per milliliter). | 4.30 (2.265) | 3.81 (1.934) | 1.97 (0.916) | 1.16 (0.426)
  Week 4: number analyzed (Participants) | 25 | 27 | 26 | 25 | 28
  Week 4 | NA (NA) — Data could not be analyzed as the values were below LLOQ (0.0977 microgram per milliliter). | 7.16 (3.290) | 2.02 (1.073) | 0.97 (0.470) | 0.85 (1.167)
  Week 8: number analyzed (Participants) | 24 | 23 | 20 | 18 | 24
  Week 8 | NA (NA) — Data could not be analyzed as the values were below LLOQ (0.0977 microgram per milliliter). | 10.54 (5.008) | 3.08 (1.806) | 1.45 (0.764) | 0.99 (0.560)
  Week 12: number analyzed (Participants) | 22 | 24 | 19 | 18 | 24
  Week 12 | NA (NA) — Data could not be analyzed as the values were below LLOQ (0.0977 microgram per milliliter). | 11.63 (5.232) | 3.10 (1.633) | 1.79 (0.836) | 0.99 (0.478)
  Week 16: number analyzed (Participants) | 20 | 22 | 14 | 14 | 23
  Week 16 | 6.84 (2.270) | 9.96 (5.107) | 3.51 (2.545) | 2.03 (1.366) | 0.98 (0.425)
  Week 20: number analyzed (Participants) | 20 | 21 | 15 | 15 | 21
  Week 20 | 9.94 (3.646) | 10.29 (4.951) | 3.92 (2.665) | 1.80 (1.030) | 1.03 (0.496)
  Week 24: number analyzed (Participants) | 18 | 17 | 14 | 13 | 19
  Week 24 | 11.04 (4.607) | 10.73 (5.182) | 3.80 (2.815) | 1.89 (1.042) | 1.04 (0.491)
  Week 24 Day 4: number analyzed (Participants) | 9 | 9 | 12 | 9 | 13
  Week 24 Day 4 | 16.46 (6.826) | 17.34 (9.046) | 9.06 (5.632) | 4.42 (1.293) | 3.36 (1.578)
  Week 24 Day 7: number analyzed (Participants) | 14 | 15 | 11 | 11 | 15
  Week 24 Day 7 | 15.14 (5.991) | 15.01 (7.853) | 9.58 (5.721) | 4.52 (1.719) | 2.80 (1.580)
  Week 26: number analyzed (Participants) | 10 | 10 | 9 | 7 | 15
  Week 26 | 10.97 (4.565) | 10.09 (6.808) | 6.49 (5.401) | 3.72 (1.434) | 1.91 (1.009)
  Week 28: number analyzed (Participants) | 16 | 15 | 13 | 14 | 19
  Week 28 | 6.93 (3.378) | 6.69 (4.329) | 4.15 (2.830) | 1.84 (0.764) | 1.06 (0.539)
  Week 30: number analyzed (Participants) | 17 | 16 | 13 | 14 | 18
  Week 30 | 4.49 (2.708) | 4.06 (2.341) | 2.42 (1.931) | 1.07 (0.529) | 0.52 (0.335)
  Week 34: number analyzed (Participants) | 14 | 16 | 14 | 12 | 17
  Week 34 | 1.88 (1.451) | 1.92 (1.403) | 0.94 (0.948) | 0.39 (0.396) | 0.10 (0.138)
  Week 38: number analyzed (Participants) | 16 | 15 | 14 | 13 | 18
  Week 38 | 0.71 (0.756) | 0.72 (0.704) | 0.29 (0.382) | 0.08 (0.114) | 0.01 (0.037)

6. Secondary Outcome: Percent Improvement From Baseline in Serum C-Reactive Protein (CRP) At Week 2 (Part A and Part B)
Description: Serum CRP is a marker of systemic inflammation. A negative change from baseline in CRP represents improvement.
Time Frame: Baseline, Week 2
Population: Population analyzed included randomized participants in Part A (excluding a site based on sponsor audit for data integrity) and Part B. Here 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Part B: Placebo | Part B: Sirukumab 100 mg q2 Weeks | Part B: Sirukumab 100 mg q4 Weeks | Part B: Sirukumab 50 mg q4 Weeks | Part B: Sirukumab 25 mg q4 Weeks | Part A: Placebo | Part A: Sirukumab 100 mg q2 Weeks
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 31 | 17 | 14
Percent change | -49.31 (246.040) | 81.46 (25.000) | 88.53 (12.675) | 85.42 (18.242) | 81.22 (24.484) | 19.97 (41.232) | 91.19 (4.812)

ADVERSE EVENTS:
Time Frame: Screening up to Week 38
Description: Safety population (SP) included all participants who received at least 1 dose of study agent (including safety data from all investigator sites irrespective of audit findings).
Groups:
- Part B - Sirukumab 25mg q4w: Participants received 25 mg of sirukumab subcutaneously every 4 weeks (q4w) for 24 weeks and in between placebo SC injections was received at Weeks 2, 6, and q4w through week 22.
Arm/Group | Part A - Placebo (Wk 0-Wk 12) | Part A - Placebo Then Sirukumab (Wk 12 to End of Study) | Part A - Sirukumab (Wk 0-Wk 12) | Part A - Sirukumab Then Placebo (Wk 12 to End of Study) | Part B - Placebo (Wk 0-Wk 12) | Part B - Placebo Then Sirukumab 100 mg q2 Weeks | Part B - Sirukumab 100mg q2w | Part B - Sirukumab 100mg q4w | Part B - Sirukumab 50mg q4w | Part B - Sirukumab 25mg q4w
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 1/17 | 0/16 | 4/30 | 2/26 | 2/30 | 5/30 | 1/30 | 3/31
Other Adverse Events (participants affected / at risk) | 12/19 | 18/18 | 12/17 | 10/16 | 15/30 | 11/26 | 20/30 | 18/30 | 25/30 | 23/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - Placebo (Wk 0-Wk 12) (N=19) | Part A - Placebo Then Sirukumab (Wk 12 to End of Study) (N=18) | Part A - Sirukumab (Wk 0-Wk 12) (N=17) | Part A - Sirukumab Then Placebo (Wk 12 to End of Study) (N=16) | Part B - Placebo (Wk 0-Wk 12) (N=30) | Part B - Placebo Then Sirukumab 100 mg q2 Weeks (N=26) | Part B - Sirukumab 100mg q2w (N=30) | Part B - Sirukumab 100mg q4w (N=30) | Part B - Sirukumab 50mg q4w (N=30) | Part B - Sirukumab 25mg q4w (N=31)
Blindness (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Arthritis Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Bursitis Infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis Staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic Inflammatory Disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Transaminases Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Facial Paresis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intracranial Aneurysm (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertebral Artery Occlusion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine Polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - Placebo (Wk 0-Wk 12) (N=19) | Part A - Placebo Then Sirukumab (Wk 12 to End of Study) (N=18) | Part A - Sirukumab (Wk 0-Wk 12) (N=17) | Part A - Sirukumab Then Placebo (Wk 12 to End of Study) (N=16) | Part B - Placebo (Wk 0-Wk 12) (N=30) | Part B - Placebo Then Sirukumab 100 mg q2 Weeks (N=26) | Part B - Sirukumab 100mg q2w (N=30) | Part B - Sirukumab 100mg q4w (N=30) | Part B - Sirukumab 50mg q4w (N=30) | Part B - Sirukumab 25mg q4w (N=31)
Haemorrhagic Diathesis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 3 | 4 | 4 | 5 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Bundle Branch Block Left (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Eye Pain (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Aphthous Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 1 | 1 | 2 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Injection Site Erythema (General disorders) | 0 | 4 | 6 | 0 | 1 | 2 | 3 | 2 | 4 | 6
Injection Site Pain (General disorders) | 1 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection Site Pruritus (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection Site Rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Injection Site Swelling (General disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection Site Urticaria (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection Site Warmth (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 2 | 1 | 0 | 0 | 5 | 0 | 1 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1
Staphylococcal Skin Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 3 | 2
Synovial Rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 4 | 2 | 0 | 1 | 1 | 4 | 7 | 10 | 6
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 1 | 3 | 4 | 6 | 3
Blood Bilirubin Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1
Blood Cholesterol Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 1
Blood Glucose Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood Insulin Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Blood Potassium Decreased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin Decreased (Investigations) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Insulin Resistance Test (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Intraocular Pressure Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2
White Blood Cell Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1 | 5 | 2 | 1 | 0 | 5 | 1 | 2 | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 0
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 3 | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 2 | 1 | 2 | 1 | 1 | 2
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 3
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.